CLINICAL TRIAL: NCT00265447
Title: Exercise and Physical Fitness for Persons With Knee Osteoarthritis: Does One Size Fit All
Brief Title: Exercise and Physical Fitness for Persons With Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H133B031120-Proj 2
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; exercise; aerobic exercise; strengthening exercise; exercise prescription; rehabilitation; physical disability; physical function; physical activity; physical fitness
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Resistance Training

ARMS (3):
- Strength training (Active Comparator): 3 months of strength training
  Interventions: Behavioral: Strength training
- Aerobic conditioning (Active Comparator): 3 months of aerobic conditioning
  Interventions: Behavioral: Aerobic conditioning
- Delayed exercise (Other): delayed exercise control group
  Interventions: Behavioral: Delayed exercise

INTERVENTIONS:
Behavioral: Strength training — 3 months of strength training
  Arms: Strength training
Behavioral: Aerobic conditioning — 3 months of aerobic conditioning
  Arms: Aerobic conditioning
Behavioral: Delayed exercise — delayed exercise control group
  Arms: Delayed exercise

SUMMARY:
The purpose of this project is to establish evidence to support specific, targeted exercise and rehabilitation recommendations for people over 50 with osteoarthritis of the knee.

DETAILED DESCRIPTION:
Physical disability and poor health often accompany knee osteoarthritis (OA), particularly as people age. This decline in function and quality of life is a complex phenomenon associated with numerous factors including pain, poor physical fitness, obesity, co-morbidity, low self-efficacy and lower extremity impairments. Furthermore, the effects of age, which have not been well studied in OA, must be considered. In addition to the functional losses associated with knee OA and aging, low levels of daily physical activity and exercise are common problems in this population for whom arthritis is a major reason for activity limitation. Evidence is accumulating that exercise can enhance health and quality of life and modify a number of the factors associated with disability. There is, however, little specific information to guide exercise prescription in the diverse population of people with knee OA. Although general benefit of exercise has been demonstrated, it is time to focus research questions on the specific types of exercise that produce specific effects; and for whom particular exercises are the most useful. Additionally, exercise has shown short term benefit, but how best to maintain gains and sustain exercise behaviors in self-directed and community settings is virtually untested. These questions are relevant to all people with knee OA, and become even more important as people grow older, become more sedentary and are at greater risk for frailty, poor health and disability.

This study is designed to: determine the efficacy of specific types of exercise by examining the effects of training on physiologic adaptations and physical performance; determine the effectiveness of a comprehensive exercise protocol performed in a supervised but non-medical setting, and describe the interaction of personal characteristics and disease severity with individual response to a particular exercise regimen.

ELIGIBILITY:
Inclusion Criteria:

community-dwelling, physician diagnosed osteoarthritis of the knee, willingness to exercise regularly, willingness to perform 3 testing sessions over a 6-month period, ability to exercise safely at a moderate level of intensity, knee osteoarthritis by clinical criteria,

WOMAC Scores as follows:

PAIN:"mild" pain on 2 items or "moderate" pain on 1 item; PHYSICAL FUNCTION: "mild" difficulty in 4 items or "moderate" difficulty in 2 items -

Exclusion Criteria:

age<50,inability to exercise and ambulate independently, physical limitation secondary to a condition that is not modifiable by exercise (e.g., active cancer), knee replacement (past or scheduled), total hip joint replacement less than 6 months ago, current participation in regular conditioning exercise, participation in another research study,

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
WOMAC Pain scale | baseline, 3 months, and 6 months
WOMAC physical function scale, muscle performance,flexibility, aerobic capacity, self-reported health status | baseline, 3 months, 6 months

SECONDARY OUTCOMES:
AIMS2 | baseline, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marian A Minor, PhD, Principal Investigator — Department of Physical Therapy, School of Health Professions, University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States